CLINICAL TRIAL: NCT07085312
Title: Evaluating the Efficacy of Exosome-Enriched Culture Media to Enhance In Vitro Maturation and Embryo Development in Poor Ovarian Responders Undergoing IVF: A Randomized Controlled Trial
Brief Title: Exosome-Enriched Culture Media to Enhance In Vitro Maturation and Embryo Development in Poor Ovarian Responders Undergoing IVF
Acronym: EXOMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertiaguerrevere (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: J-298384255-2
Record Dates: First submitted 2025-07-07; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Poor Ovarian Response; Female Infertility of Other Origin; Oocyte Immaturity
Keywords: exosomes; in vitro maturation; oocyte maturation; IVF; poor ovarian responders

STUDY DESIGN:
Masking Description: "Not applicable. No additional parties are masked in this trial."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian Stimulation with MI Oocyte Allocation to Exosome vs. Standard Media (Experimental): All participants undergo controlled ovarian stimulation and oocyte retrieval following a standard antagonist protocol. Retrieved MI oocytes from each patient are then allocated to two different in vitro culture conditions: (1) standard IVF media, and (2) IVF media supplemented with 10 µg of GMP-certified exosomes per well. This design allows within-patient comparison of oocyte maturation, fertilization, and embryo development outcomes under the two culture environments.
  Interventions: Procedure: Exosome-Enriched IVF Culture

INTERVENTIONS:
Procedure: Exosome-Enriched IVF Culture — IVF culture media supplemented with 10 µg per well of GMP-certified exosomes (Exosmart or equivalent). Retrieved MI oocytes are cultured in this media for up to 4 hours to assess progression to MII.

SUMMARY:
Evaluating the Efficacy of Exosome-Enriched Culture Media to Enhance In Vitro Maturation and Embryo Development in Poor Ovarian Responders Undergoing IVF

Summary:

This is a prospective, randomized controlled trial designed to assess whether supplementing standard IVF culture media with exosomes can improve the short-term in vitro maturation (IVM) of immature MI oocytes in poor ovarian responder patients.

Sixty women aged 35-42 who meet Bologna criteria for poor ovarian response will be recruited and randomized into two groups:

Control group: MI oocytes cultured in standard IVF media.

Intervention group: MI oocytes cultured in IVF media supplemented with 10 µg of GMP-certified exosomes per well.

The primary outcome is the proportion of MI oocytes maturing to MII within 4 hours. Secondary outcomes include fertilization rates, embryo quality, blastocyst development, and clinical pregnancy rates.

This study aims to explore a novel approach to improving oocyte yield and embryo development in poor responder IVF cycles, potentially reducing the need for repeated treatments and enhancing patient outcomes.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial designed to evaluate the efficacy of exosome-enriched culture media in promoting the short-term in vitro maturation (IVM) of immature oocytes retrieved from poor ovarian responder patients undergoing in vitro fertilization (IVF).

Rationale:

Poor ovarian responders represent a significant clinical challenge in assisted reproductive technology (ART), often yielding a low number of mature metaphase II (MII) oocytes after controlled ovarian stimulation. A substantial proportion of oocytes retrieved in these patients remain at the metaphase I (MI) stage and traditionally show limited capacity for maturation, thereby reducing the pool of oocytes available for fertilization.

Emerging preclinical data and our pilot observations suggest that exosomes-extracellular vesicles containing bioactive molecules such as miRNAs, proteins, and growth factors-play a crucial role in follicular development and may facilitate oocyte meiotic progression. Incorporating exosomes into IVF culture media could therefore represent a novel strategy to enhance in vitro maturation of MI oocytes and improve outcomes in this difficult-to-treat population.

Study Design and Methods:

The study will enroll 60 women aged 35 to 42 years, all meeting at least two Bologna criteria for poor ovarian response. Patients will undergo controlled ovarian stimulation with antagonist protocols and oocyte retrieval approximately 36-37 hours after hCG administration. Retrieved oocytes will be classified as MI or MII.

MI oocytes will be randomized on a per-patient basis into two groups:

Control group: MI oocytes cultured in pre-equilibrated Cook IVF media without additional supplementation.

Intervention group: MI oocytes cultured in the same media supplemented with 10 µg/well of GMP-certified exosomes (sourced from Exosmart or an equivalent validated supplier).

Oocytes will be monitored for progression from MI to MII at intervals up to 4 hours. Subsequent ICSI will be performed on matured oocytes, and resulting embryos will be cultured to blastocyst stage following standard laboratory protocols.

Outcomes:

The primary endpoint is the proportion of MI oocytes achieving maturation to MII within 4 hours of culture.

Secondary endpoints include fertilization rates (2PN formation), day 3 and blastocyst morphological grading, implantation rates, and clinical pregnancy rates per embryo transfer.

Statistical Considerations:

Data will be analyzed using chi-square or Fisher's exact tests for categorical variables such as maturation and fertilization rates. Logistic regression may be used to adjust for confounding factors such as patient age, baseline AMH, and gonadotropin dose. A p-value <0.05 will be considered statistically significant.

Ethical Considerations:

All patients will provide written informed consent before participation. The study will be conducted in compliance with the Declaration of Helsinki, local regulations, and Good Clinical Practice (GCP) guidelines. The protocol will be reviewed and approved by the appropriate Institutional Review Board (IRB) prior to initiation.

Potential Impact:

By investigating the role of exosome supplementation in improving the maturation of MI oocytes, this study seeks to expand the pool of usable oocytes in poor responder IVF cycles. This could translate to higher embryo availability, reduced cycle cancellations, and ultimately improved pregnancy outcomes in a patient group historically characterized by low success rates.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

Women aged 35 to 42 years

Undergoing IVF with an antagonist protocol

Meet at least two Bologna criteria for poor ovarian response

Provide written informed consent -

Exclusion Criteria:

* Exclusion Criteria:

Severe male factor infertility requiring surgical sperm retrieval

Known untreated hydrosalpinx

Uterine anomalies that impair implantation

Known chromosomal abnormalities

Participation in another investigational study within 3 months

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female, Self-identified women.
Enrollment: 10 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Proportion of MI Oocytes Achieving MII Maturation | Within 4 hours post-culture
  The primary outcome is the percentage of retrieved MI oocytes that progress to MII after 2-4 hours of culture in exosome-enriched versus standard IVF media. Oocyte maturation is assessed morphologically under an inverted microscope.

SECONDARY OUTCOMES:
Fertilization Rate | 18-20 hours post-ICSI
  Percentage of matured MII oocytes that exhibit normal 2PN fertilization after ICSI.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertiaguerrevere Fertility, Caracas, Distrito Federal, Venezuela

IPD SHARING:
Plan to Share IPD: No
"Individual participant data (IPD) will not be shared due to the small sample size, the sensitive nature of reproductive and embryology data, and to protect patient confidentiality in this specialized cohort. Future larger studies may consider data sharing agreements under appropriate anonymization and ethical safeguards."

REFERENCES:
- [Result] Song J, Guo X, Zhang B, Zhang Q, Han Y, Cao D, Yao Y. Human Umbilical Cord Mesenchymal Stem Cells Derived Exosomes Improved The Aged Mouse IVM Oocytes Quality. Reprod Sci. 2024 Sep;31(9):2808-2819. doi: 10.1007/s43032-024-01566-z. Epub 2024 Apr 30. PMID 38689080
- [Result] Melo P, Navarro C, Jones C, Coward K, Coleman L. The use of autologous platelet-rich plasma (PRP) versus no intervention in women with low ovarian reserve undergoing fertility treatment: a non-randomized interventional study. J Assist Reprod Genet. 2020 Apr;37(4):855-863. doi: 10.1007/s10815-020-01710-z. Epub 2020 Feb 7. PMID 32030554

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT07085312/Prot_SAP_ICF_000.pdf